CLINICAL TRIAL: NCT06948903
Title: Investigation of the Relationship Between Central Sensitization Symptoms and Cognitive Dysfunction in Patients With Fibromyalgia
Brief Title: Relationship Between Central Sensitization Symptoms and Cognitive Dysfunction in Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 11111
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia; Cognitive Dysfunction; Central Sensitisation
Keywords: Fibromyalgia; Cognitive Dysfunction; Central Sensitisation
MeSH Terms: conditions — Fibromyalgia; Cognitive Dysfunction | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with fibromyalgia
  Interventions: Diagnostic Test: Central Sensitization Inventory; Diagnostic Test: The Montreal Cognitive Assessment; Diagnostic Test: Cognitive Symptom Severity Scale-Extended; Other: Fibromyalgia Impact Questionnaire; Other: Numeric rating scale; Other: Hospital Anxiety and Depression Scale

INTERVENTIONS:
Diagnostic Test: Central Sensitization Inventory — The Central Sensitization Inventory is used by some researchers to investigate pain sensitivity through symptoms associated with central sensitization and related comorbidities. It can help determine the severity of central sensitization. The scale was developed to detect central sensitization in patients with chronic pain and consists of two sections: Section A and Section B. For scoring purposes, only Section A is used. A score of 40 or higher out of 100 is associated with an increased likelihood of central sensitization.
Diagnostic Test: The Montreal Cognitive Assessment — The Montreal Cognitive Assessment was initially developed as a test for mild cognitive impairment, but has also been determined to match qualities of the mini mental state examination 80. It assesses seven areas of cognition for a total possible score of 30 points. A score of 21 or less is indicative of cognitive impairment in Turkish population.
Diagnostic Test: Cognitive Symptom Severity Scale-Extended — The Cognitive Symptom Severity Scale extends the scale of the original cognitive symptom severity scale. Participants are asked to rate their cognitive symptoms related to concentration and memory on a single scale ranging from 1-5, rather than the original 1-3, where higher scores indicate greater severity.
Other: Fibromyalgia Impact Questionnaire — The Fibromyalgia Impact Questionnaire is composed of 10 items. The first item contains 11 questions related to physical functioning - each question is rated on a 4 point Likert type scale. Items 2 and 3 ask the patient to mark the number of days they felt well and the number of days they were unable to work (including housework) because of fibromyalgia symptoms. Items 4 through 10 are horizontal linear scales marked in 10 increments on which the patient rates work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety and depression. The maximum scale score is 100, with higher scores associated with increasing disability.
Other: Numeric rating scale — Numeric Rating Scale will be used to determine pain intensity during assessments. Participants will be asked to rate their pain intensity by selecting a value between 0 and 10. Higher scores are associated with increased pain severity.
Other: Hospital Anxiety and Depression Scale — This scale is used to assess anxiety and depression symptoms and consists of 14 items (7 items for anxiety, 7 items for depression). For each subscale, scores range from 0 to 21: • 0-7 points: No symptoms or very mild symptoms • 8-10 points: Moderate symptoms • 11 points or higher

SUMMARY:
The aim of the study is to investigate the relationship between central sensitization parameters and cognitive dysfunction in patients with fibromyalgia.The main questions it aims to answer are:

Do central sensitization symptoms affect cognitive dysfunction in patients with fibromyalgia? To what extent do central sensitization symptoms affect objective and subjective cognitive complaints in fibromyalgia patients? How do cognitive complaints relate to other clinical parameters, including disease severity, in these patients?

DETAILED DESCRIPTION:
Central sensitization is defined as an increase in pain sensitivity with amplification of neuron-derived signals in the central nervous system. Fibromyalgia is a disease characterized by chronic widespread pain, and although its etiology and pathophysiology are still not fully known, it is considered a major member of the group of diseases known as central sensitivity syndromes, which progress with impaired pain regulation.

Fibromyalgia negatively affects the patient's functionality in various ways. One of these is cognitive dysfunction, and previous studies have shown that fibromyalgia patients experience significant deterioration in all parameters related to cognitive function compared to healthy controls. Central sensitization has been shown to be associated with comorbidities such as depression, anxiety, sleep disorders and fatigue in many disease groups, including fibromyalgia, and data on its effect on cognitive dysfunction are limited.

A study found that impaired conditioned pain modulation, one of the methods used in the evaluation of central sensitization in fibromyalgia patients, was associated with cognitive dysfunction.In addition, cognitive impairment in these patients is associated with a decrease in the quality of life of the patients and is suggested to be one of the important clinical findings of the disease. Considering all these data, it seems likely that central sensitization negatively affects cognitive function in fibromyalgia, and this study aimed to examine in detail the relationship between central sensitization and cognitive dysfunction in fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with fibromyalgia according to American College of Rheumatology 2016 criteria
* Being between 18-65 years old
* Being literate
* Accepting to participate in the study

Exclusion Criteria:

* Concomitant systemic inflammatory disease, central nervous system disease (cortical involvement), active infection and malignancy history
* History of illness that may lead to cognitive impairment
* Being <18 and >65 years old
* Being illiterate
* Not accepting to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Fibromyalgia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Central Sensitization Inventory | 6 months
  The Central Sensitization Inventory is used by some researchers to investigate pain sensitivity through symptoms associated with central sensitization and related comorbidities. It can help determine the severity of central sensitization. The scale was developed to detect central sensitization in patients with chronic pain and consists of two sections: Section A and Section B. For scoring purposes, only Section A is used. A score of 40 or higher out of 100 is associated with an increased likelihood of central sensitization.
Montreal Cognitive Assessment | 6 months
  The Montreal Cognitive Assessment was initially developed as a test for mild cognitive impairment, but has also been determined to match qualities of the mini mental state examination 80. It assesses seven areas of cognition for a total possible score of 30 points. A score of 21 or less is indicative of cognitive impairment in Turkish population.

SECONDARY OUTCOMES:
Cognitive Symptom Severity Scale-Extended | 6 months
  The Cognitive Symptom Severity Scale extends the scale of the original cognitive symptom severity scale. Participants are asked to rate their cognitive symptoms related to concentration and memory on a single scale ranging from 1-5, rather than the original 1-3, where higher scores indicate greater severity.
Fibromyalgia Impact Questionnaire | 6 months
  This scale is composed of 10 items. The first item contains 11 questions related to physical functioning - each question is rated on a 4 point Likert type scale. Items 2 and 3 ask the patient to mark the number of days they felt well and the number of days they were unable to work (including housework) because of fibromyalgia symptoms. Items 4 through 10 are horizontal linear scales marked in 10 increments on which the patient rates work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety and depression. The maximum scale score is 100, with higher scores associated with increasing disability.
Hospital Anxiety and Depression Scale | 6 months
  This scale is used to assess anxiety and depression symptoms and consists of 14 items (7 items for anxiety, 7 items for depression). For each subscale, scores range from 0 to 21: • 0-7 points: No symptoms or very mild symptoms • 8-10 points: Moderate symptoms • 11 points or higher
Numeric rating scale | 6 months
  Numeric Rating Scale will be used to determine pain intensity during assessments. Participants will be asked to rate their pain intensity by selecting a value between 0 and 10. Higher scores are associated with increased pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Yücel, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Health Sciences University, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data sharing not planned

REFERENCES:
- [Result] Akinci A, Al Shaker M, Chang MH, Cheung CW, Danilov A, Jose Duenas H, Kim YC, Guillen R, Tassanawipas W, Treuer T, Wang Y. Predictive factors and clinical biomarkers for treatment in patients with chronic pain caused by osteoarthritis with a central sensitisation component. Int J Clin Pract. 2016 Jan;70(1):31-44. doi: 10.1111/ijcp.12749. Epub 2015 Nov 11. PMID 26558538
- [Result] Bell T, Trost Z, Buelow MT, Clay O, Younger J, Moore D, Crowe M. Meta-analysis of cognitive performance in fibromyalgia. J Clin Exp Neuropsychol. 2018 Sep;40(7):698-714. doi: 10.1080/13803395.2017.1422699. Epub 2018 Feb 1. PMID 29388512
- [Result] Coppieters I, Ickmans K, Cagnie B, Nijs J, De Pauw R, Noten S, Meeus M. Cognitive Performance Is Related to Central Sensitization and Health-related Quality of Life in Patients with Chronic Whiplash-Associated Disorders and Fibromyalgia. Pain Physician. 2015 May-Jun;18(3):E389-401. PMID 26000686
- [Result] Bertolucci PH, de Oliveira FF. Cognitive impairment in fibromyalgia. Curr Pain Headache Rep. 2013 Jul;17(7):344. doi: 10.1007/s11916-013-0344-9. PMID 23709236
- [Result] Elkana O, Yaalon C, Raev S, Sobol N, Ablin JN, Shorer R, Aloush V. A modified version of the 2016 ACR fibromyalgia criteria cognitive items results in stronger correlations between subjective and objective measures of cognitive impairment. Clin Exp Rheumatol. 2021 May-Jun;39 Suppl 130(3):66-71. doi: 10.55563/clinexprheumatol/403mpp. Epub 2021 Mar 16. PMID 33734966
- [Result] Duzce Keles E, Birtane M, Ekuklu G, Kilincer C, Caliyurt O, Tastekin N, Is EE, Ketenci A, Neblett R. Validity and reliability of the Turkish version of the central sensitization inventory. Arch Rheumatol. 2021 Oct 18;36(4):518-526. doi: 10.46497/ArchRheumatol.2022.8665. eCollection 2021 Dec. PMID 35382371
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Kaya Y, Aki OE, Can UA, Derle E, Kibaroglu S, Barak A. Validation of Montreal Cognitive Assessment and Discriminant Power of Montreal Cognitive Assessment Subtests in Patients With Mild Cognitive Impairment and Alzheimer Dementia in Turkish Population. J Geriatr Psychiatry Neurol. 2014 Jun;27(2):103-9. doi: 10.1177/0891988714522701. Epub 2014 Feb 26. PMID 24578463
- [Result] Sarmer S, Ergin S, Yavuzer G. The validity and reliability of the Turkish version of the Fibromyalgia Impact Questionnaire. Rheumatol Int. 2000 Dec;20(1):9-12. doi: 10.1007/s002960000077. PMID 11149662